CLINICAL TRIAL: NCT00436683
Title: An Open Label, Dose-Ranging Study to Establish the Tolerability of Magnesium Iron Hydroxycarbonate in Haemodialysis Subjects With Hyperphosphataemia.
Brief Title: Dose Ranging Study of Magnesium Iron Hydroxycarbonate in Haemodialysis Subjects With Hyperphosphataemia
Acronym: ACT3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ineos Healthcare Limited (Industry)
Responsible Party: Chief Medical Officer, INEOS Healthcare Limited
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IH 003 (ACT3)
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2009-08-10 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Kidney Failure
Keywords: Hyperphosphataemia; Phosphate binder
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperphosphatemia | interventions — iron-magnesium hydroxycarbonate; Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Dose titration on active
  Interventions: Drug: Fermagate
- 2 (Active Comparator): Dose titration
  Interventions: Drug: Sevelamer HCl

INTERVENTIONS:
Drug: Fermagate — Film coated tablet 500mg
  Other Names: Alpharen
  Arms: 1
Drug: Sevelamer HCl — tablet 800mg
  Other Names: RenaGel
  Arms: 2

SUMMARY:
Magnesium iron hydroxycarbonate is a phosphate binder that absorbs phosphate from food, reducing the amount that the body can absorb.

The purpose of this study is to determine how well a range of different doses of fermagate are tolerated by the subjects in the trial.

DETAILED DESCRIPTION:
High levels of phosphate in the blood are linked with serious effects, due to calcium imbalances (high levels of parathyroid hormone (PTH), bone disease, formation of calcium deposits in the body, and blood-vessel disease.

Current guidelines indicate that blood phosphorus levels should be maintained between 1.13 to 1.78 mmol/L in patients who receive hemodialysis.

The purpose of this study is to determine the range of dosages which are tolerated by patients with hyperphosphatemia, undergoing haemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects on active haemodialysis, aged 18 years or over who are able to comply with study procedures
* Written informed consent given
* On a stable haemodialysis regimen (three times per week) for at least 3 months and be unlikely to change their dialysis prescription during the study period
* On a stable dose of phosphate binder for at least 1 month prior to screening
* Willing to abstain from taking any phosphate binder or oral magnesium-, aluminium- or iron-containing products and preparations, other than the study medication
* Willing to avoid any intentional changes in diet such as fasting, dieting or overeating
* On a dialysate magnesium ion concentration of ≤1.0 mmol/L for at least 1 month prior to screening

Exclusion Criteria:

* Received a cardiac transplant
* Heart failure according to New York Heart Association (NYHA) Functional IV Classification
* Participation in any other clinical trial using an investigational product or device within the previous 4 weeks
* A significant history of alcohol, drug or solvent abuse in the opinion of the investigator
* Any disease or condition, physical or psychological, which in the opinion of the investigator would compromise the safety of the subject or increase the likelihood of the subject being withdrawn
* Clinically significant laboratory findings (at screening for this subject population) in the opinion of the investigator
* Any history of recent clinically significant malignancy
* A significant illness (excluding renal disease) in the 4 weeks before screening
* A history of poorly controlled epilepsy
* Female subjects who are lactating or pregnant. Women of childbearing potential (pre-menopausal and not surgically sterilised) unless they are using a reliable contraceptive method, that is, barrier methods, hormones or intrauterine device
* Allergy to magnesium iron hydroxycarbonate or sevelamer or any component of the formulations
* Any condition that affects the reliability of measuring QT interval, for example, an irregular heart rhythm such as atrial fibrillation or frequent ectopic activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-02; Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Assessment of intolerance | 10 weeks

SECONDARY OUTCOMES:
Assessment of QTc interval | 10 weeks
Change from baseline in serum electrolytes | 10 weeks
Change from baseline in parathyroid hormone (PTH) | 10 weeks
Reduction of serum magnesium removal during dialysis | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Taal, MBChB MD FRCP, Principal Investigator — Derby City Hospital
Locations (15):
- United Kingdom (15):
  - Department of Renal Medicine, Derby City General Hospital, Uttoxeter Road, Derby, Derbyshire
  - Queens Dialysis Unit, Rom Valley Way, Romford, Essex
  - Renal Unit, Queen Elizabeth Hospital, Edgbaston, Birmingham
  - Ash Haemodialysis Unit, Hospital of St Cross, University Hospital of Coventry & Warwickshire NHS Trust, Clifford Bridge Road, Coventry
  - Haemodyialysis unit, Department of Nephrology, Walsgrave Hospital, University of Coventry & Warwickshire NHS Trust, Clifford Bridge Road, Coventry
  - Renal Dialysis Unit, Western Infirmary, Dumbarton Road, Glasgow
  - Renal Dialysis Unit, Gartnavel General Hospital, Glasgow
  - Renal Unit, The Royal London Hospital, Whitechapel, London
  - Whipps Cross Renal Unit, Whipps Cross University Hospital, Whipps Cross Road, Leytonstone, London
  - Wanstead Renal Unit, 29 Cambridge Park, Wanstead, London
  - Renal Unit, St Bartholomew's Hospital, West Smithfield, London
  - Central Manchester & Manchester Childrens Hospital NHS Trust, Renal Dialysis Unit, Manchester Royal Infirmary, Oxford Rd, Manchester
  - Central Manchester & Manchester Childrens Hospital NHS Trust, Renal Dialysis Unit, Wythenshawe Hospital, Southmoor Rd, Manchester
  - Haemodialysis Unit, Royal Berkshire Hospital, Royal Berkshire Hospital, Royal Berkshire NHS Foundation Trust, London Rd, Reading
  - Renal Services, Hope Hospital, Salford

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086